CLINICAL TRIAL: NCT00387777
Title: Multiple Dose Bioequivalence Trial Comparing a New Analgesic Transdermal Patch Formulation to an Analgesic Reference Patch.
Brief Title: Multiple Dose Trial Comparing the Plasma Levels of Two Different Analgesic Transdermal Patch Formulations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 631766; 2006-003177-27 (EudraCT Number); HP5303/10 (Other: Grünenthal GmbH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Buprenorphine; Transdermal patch; multidose; Centrally acting analgesic; Plasma level; Healthy volunteers
MeSH Terms: interventions — Transdermal Patch; prolyl-proline; Buprenorphine

INTERVENTIONS:
Drug: Patch with centrally acting analgesic
Drug: Transtec(R) PRO (buprenorphine)

SUMMARY:
The purpose of this study is to determine whether Transtec(R) PRO 70 µg/h and a new buprenorphine patch formulation lead to same plasma levels of buprenorphine after multiple dose application.

DETAILED DESCRIPTION:
Main: To demonstrate the bioequivalence of the new buprenorphine transdermal patch T2rev formulation containing 13 mg buprenorphine (Test) as compared to Transtec(R) PRO 70 µg/h patch transdermal patch containing 40 mg buprenorphine as reference after multiple patch application. Pharmacokinetic target parameters are AUCss,Tau and Css,max.

Further: To assess the safety, tolerability, skin tolerability and adhesiveness of the patch applications. To evaluate the following further Pharmacokinetic parameters: Css,min, Css,ave, PTF, Swing, tss,max, and t1/2,z

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian subjects, aged 18 - 55 years
* BMI between 18 and 30 kg/m2 inclusive, with a lover limit of body weight of 50 kg
* Subjects must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters
* Subjects giving written informed consent to participate within this trial

Exclusion Criteria:

* Resting pulse rate <= 45 or >= 100 beats/min
* Resting blood pressure:systolic blood pressure <= 90 and >= 160 mmHg, diastolic blood pressure <= 40 and >= 100 mmHg
* History or presence of orthostatic hypotension
* Positive test of HIV type 1/2 antibodies, HBs antigen, HBc antibodies, HCV antibodies
* Participation in another clinical trial in the last 30 days before starting this trial (i.e., first administration of IMP)
* Positive drug of abuse screening
* Diseases or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* Marked repolarisation abnormality (e.g., suspicious or definite congenital long QT syndrome with QT/QTc>500msec or prolonged QTc, i.e.>450msec) or co-medication that is known to influence cardiac repolarisation substantially
* Bronchial asthma
* Definite or suspected history of drug allergy or hypersensitivity
* Subjects who have received any prescribed and non-prescribed systemic or topical medication like analgesics, NSAIDs (except standard dose of a NSAID once a week for the treatment of headache), hypnotics, sedatives, narcotics, neuroleptics or other medications that may lower the seizure threshold, MAO-inhibitors, serotonin-reuptake-inhibitors, tricyclic antidepressants, other centrally acting substances and substances which are known to interact with the drug metabolizing enzymes (e.g., inhibitors or inducers of CYP3A4 or CYP2D6) four weeks prior to the start of the trial (i.e, first administration of IMP). Each case has to be decided upon individually by the investigator after consultation with the sponsor
* Evidence of alcohol or drug abuse
* Not able to abstain from consumption of:
* Caffeine containing beverages or food (tea, coffee, cola, chocolate, etc.)
* Quinine containing beverages or food (bitter lemon, tonic water)
* Grapefruit juice (sweet, sour)
* Poppy seeds containing beverages or food
* Blood loss (> 100 mL) due to e.g., blood donation within 3 months before starting this trial (i.e., first administration of IMP)
* History of seizures or at risk (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness)
* Known or suspected of not being able to comply with the trial protocol
* Not able to communicate meaningfully with the investigator and staff
* Smoking of > 10 cigarettes/day or equivalent.

Trial specific exclusion criteria:

* Subjects not able to abstain from strenuous exercise during the whole course of the trial
* Abnormality (e. g. scar, tattoo) or unhealthy skin at application site according to examination by the investigator
* Existing chronic skin disease or history of skin disease at the application site within the last 4 weeks
* Presence of one of the contraindications as detailed in the current Summary of Product Characteristics (SmPC).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Baumann-Noss, MD, Principal Investigator — IKP Mannheim
Locations (1):
- IKP, Mannheim, Germany